CLINICAL TRIAL: NCT00720148
Title: Phase IB Dose Escalation Study of Bortezomib (VELCADE) Administered Weekly for 4 Weeks and Sunitinib (SU-011248) Administered Daily for 4 Weeks Followed by a 14 Day Rest in Patients With Refractory Solid Tumors
Brief Title: A Phase I Trial of Bortezomib and Sunitinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Pfizer (Industry)
Responsible Party: Principal Investigator, R. Donald Harvey, PharmD, PharmD, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00003549; 3549 (Other: Other)
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Solid Tumors
Keywords: Solid tumors
MeSH Terms: interventions — Sunitinib; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sunitinib and Bortezomib — 50 mg/m2, IV (in the vein)on day 5 of each 28 day cycle. Number of cycles: until progression or unacceptable toxicity develops
  Other Names: Sutent; Velcade

SUMMARY:
The purpose of this study is to test the effect of the combination of sunitinib and bortezomib. We will see what effects it has on your cancer and find the highest dose of each agent that can be given without causing severe side effects.

DETAILED DESCRIPTION:
This is a Phase I study assessing the combination of bortezomib and sunitinib in patients with solid tumors that are refractory to standard chemotherapy.

The study will take place in two stages. In both stages, patients will receive sunitinib orally with food once daily for 4 weeks and bortezomib by injection into a vein once a week for 4 weeks. This will be followed by 2 weeks of rest. This 6-week period is called one cycle.

In stage 1, a maximum of 10 patients will be treated sequentially with increasing doses of sunitinib (and a fixed dose of bortezomib). Each dose level must be well tolerated for the next patient to start treatment at the next dose level. Whichever is the highest dose of sunitinib that is well tolerated will then be used for the next stage.

In stage 2, a maximum of 20 patients will be treated sequentially with increasing doses of bortezomib (and a fixed dose of sunitinib). Each dose level must be well tolerated for the next patient to start treatment at the next dose level.

Together, the two stages will determine the highest doses of both sunitinib and bortezomib that are well tolerated when given this combination. Determining these optimal doses is the primary aim of this study. Patients will also be followed to see whether their tumor responds to the treatment.

If a patient's cancer remains stable or improves, they can repeat the treatment cycles. There is no defined end date to this study since patients will be followed for the duration of their survival.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Refractory advanced solid tumor that has failed standard therapy.
* ECOG PS ≤ 2
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.
* Cardiac ejection fraction is more than 45%

Exclusion Criteria:

* Patient has a platelet count of <100 x 109/L within 14 days before enrollment.
* Patient has an absolute neutrophil count of ANC <1.0 x 109/L within 14 days before enrollment.
* Patient has a calculated or measured creatinine clearance of <30 mL/minute within 14 days before enrollment.
* AST, ALT, total bilirubin > twice the upper limits of normal.
* Received radiation to more than 30% of marrow volume
* Patient has greater than or equal to Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to sunitinib, bortezomib, boron or mannitol.
* Uncontrolled hypertension
* History of venous thromboembolic events.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum Beta-human chorionic gonadotropin (Beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Hemorrhagic tendency of the tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity of combination therapy with sunitinib and bortezomib | every week

SECONDARY OUTCOMES:
Tumor shrinkage | every 6 weeks while on treatment

CONTACTS AND LOCATIONS:
Overall Officials: John Kauh, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States